CLINICAL TRIAL: NCT02442570
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled, Exploratory, Dose-ranging Study to Evaluate the Safety, Effectiveness and Pharmacokinetics of Three Courses of DC-TAB Treatment in Patients With Multiple Sclerosis
Brief Title: A Study to Evaluate Safety and Efficacy of DC-TAB in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Delta Crystallon BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DC-002
Record Dates: First submitted 2015-05-01; First posted 2015-05-13 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis
Keywords: alpha B-crystallin; immune tolerance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DC-TAB 7.5 mg (Active Comparator): three intravenous injections of 7.5 mg DC-TAB (recombinant human alpha B-crystallin), 2 months apart
  Interventions: Biological: recombinant human alpha B-crystallin
- DC-TAB 12.5 mg (Active Comparator): three intravenous injections of 12.5 mg DC-TAB (recombinant human alpha B-crystallin), 2 months apart
  Interventions: Biological: recombinant human alpha B-crystallin
- DC-TAB 17.5 mg (Active Comparator): three intravenous injections of 17.5 mg DC-TAB (recombinant human alpha B-crystallin), 2 months apart
  Interventions: Biological: recombinant human alpha B-crystallin
- placebo (Placebo Comparator): three intravenous injections of placebo, 2 months apart
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Biological: recombinant human alpha B-crystallin — intravenous injections
  Other Names: HspB5; CRYAB; DC-TAB
  Arms: DC-TAB 12.5 mg; DC-TAB 17.5 mg; DC-TAB 7.5 mg
Other: Placebo comparator — intravenous injection
  Other Names: phosphate-buffered saline
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate safety and clinical efficacy of DC-TAB in multiple sclerosis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, exploratory, dose-ranging Phase IIa study in multiple sclerosis patients to evaluate the safety, tolerability, T-cell tolerance inducing effect, clinical effects and pharmacokinetics of intravenous DC-TAB, a solution of recombinant human alpha B-crystallin.

At entry, patients were randomized to one of the treatments, placebo, 7.5 mg DC-TAB, 12.5 mg DC-TAB or 17.5 mg DC-TAB in a 1:1:1:1 fashion. Patients received a single intravenous bolus injection which was repeated twice with 2-month intervals during the 6-month monitoring period. The goal of such injection was to induce antigen-specific T-cell tolerance. The study consisted of two parts, a treatment period of 24 weeks, and a follow-up period of an additional 24 weeks. Patients returned to the hospital weekly during the first month, and monthly thereafter.

The primary analysis was performed on data collected in the treatment period, and was performed after all patients had completed 24 weeks into the study. An additional analysis was performed once all patients had completed the full 48 weeks of the study. Patients and site study personnel remained blinded throughout the study.

After 12 and 24 patients completed 4 weeks into the study, and after 24 patients had completed 12 weeks of follow-up, a partially blinded safety review was conducted by an independent drug safety monitoring board to verify safety of the intervention in MS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite relapsing multiple sclerosis, according to the McDonald criteria
2. Abnormal MRI consistent with MS
3. Neurologically stable for at least one month
4. At least one clinical relapse over the previous year, or two relapses over the past two years, or one or more gadolinium-enhancing MRI lesion(s) at the time of screening.
5. An EDSS score less than 6
6. Body weight less than 130 kg
7. Use of adequate and stable contraception for 3 months prior to study initiation, during the course of the study and 30 days thereafter or must have undergone clinically documented total hysterectomy and/or oophorectomy, surgical sterilization, or be postmenopausal defined by amenorrhea for at least 12 months and confirmed with a FSH greater than 40 mIU/mL.
8. If patients claim abstinence as their method of contraception, they must be willing to agree to use condoms if they became sexually active from 14 days prior to the first dose of the study drug through 90 days beyond the conclusion of the study.
9. Being informed of the nature and aims of the study, and having given written consent to participate in this study in accordance with local laws and requirements
10. Being willing to comply with the protocol, and understand the information given, and the text of the consent form

Exclusion Criteria:

1. Primary progressive multiple sclerosis
2. Use of systemic corticosteroid treatment for more than 3 days within 30 days prior to screening
3. Plasmapheresis, or intravenous gammaglobulins less than 2 months before screening
4. Treatment with natalizumab less than one year before screening
5. Previous immunosuppressive treatment
6. Previous treatment with any leukocyte-targeting monoclonal antibody
7. Previous treatment with oral immune-modulatory agents (cladribine, fingolimod, laquinimod, fumarate)
8. Pregnant women, women planning to become pregnant and breastfeeding women
9. A history of or currently active clinically significant cardiac (including clinically significant ECG abnormalities in the opinion of the PI), pulmonary, gastrointestinal, hepatic, renal, pancreatic, or neurological disease
10. ALT, AST and/or gamma-GT above 3 times the upper limit of normal
11. Serum creatinine above 1.5 times the upper limit of normal or an eGFR < 60 mL/min/1.73 m2
12. Hemoglobin < 7.0 mmol/l for females and < 8 mmol/l for males; leukocytes > 20*109/l or < 3.5*109/l; platelets < 125*109/l
13. SBP > 160 mmHg and/or DBP > 100 mmHg
14. Acute respiratory or other active infections
15. Fever (body temperature > 38.0 °C on day 1)
16. Blood donation or significant blood loss within 90 days of first study medication dosing
17. Plasma donation within 7 days of first study medication dosing
18. Having received blood or blood products in the last 6 months
19. Participation in another clinical study within 90 days of the start of this trial or planning participation in another clinical trial during this study or in the 4 weeks after last visit
20. Taking anti-coagulation or anti-platelet medication with the exception of NSAID's.
21. History of drug addiction (positive drug screen) or excessive use of alcohol (weekly intake more than 28 units of alcohol), or psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the patient to comply with the protocol requirements
22. Vaccination with any vaccine within 4 weeks prior to dosing of the study medication
23. History of serious adverse reactions or hypersensitivity to any medicinal product
24. History of a malignancy other than skin cell basalioma 5 years prior to screening
25. Any physical condition that would, in the opinion of the investigator, place the patient at an unacceptable health risk or risk of injury or render the patient unable to meet the requirements of the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 48 weeks
  Frequency of adverse events

SECONDARY OUTCOMES:
Tolerability (Injection site abnormalities) | 48 weeks
  Injection site abnormalities
Clinical efficacy (Number of Gadolinium-enhancing MRI lesions) | 48 weeks
  Number of Gadolinium-enhancing MRI lesions
Pharmacokinetics (serum levels of DC-TAB) | 8 hours
  Serum levels of DC-TAB
Antigen-specific T-cell response | 48 weeks
  Strength of antigen-specific T cell responses
Antibody response | 48 weeks
  Serum levels of anti-DC-TAB antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Lilly Boneva, MSc, Study Director — Population Services International
Locations (5):
- Bulgaria (5):
  - Sveti Naum Hospital, Sofia
  - National Cardiology Hopsital, Sofia
  - Tokuda Hospital Sofia, Sofia
  - Aleksandrovska Hospital, Sofia
  - Military Medical Academy, Sofia

REFERENCES:
- [Derived] van Noort JM, Bsibsi M, Nacken PJ, Verbeek R, Venneker EH. Therapeutic Intervention in Multiple Sclerosis with Alpha B-Crystallin: A Randomized Controlled Phase IIa Trial. PLoS One. 2015 Nov 23;10(11):e0143366. doi: 10.1371/journal.pone.0143366. eCollection 2015. PMID 26599332